CLINICAL TRIAL: NCT07325864
Title: Molecular Phenotyping of Primitive Lung Cancer and Metastatic Site
Status: Recruiting | Type: Observational
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: UID 4058; IEO 1956 (Other: Comitato Etico degli IRCCS Istituto Europeo di Oncologia e Centro Cardiologico Monzino)
Record Dates: First submitted 2025-12-23; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: NSCLC; Lung Cancer (Diagnosis)
Keywords: lung cancer; nsclc; NGS; pleural metastasis; oligometastatic
MeSH Terms: conditions — Lung Neoplasms; Disease; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Molecular Phenotyping of Primitive Lung Cancer and Metastatic Site in patient diagnosed with NSCLC: To investigate the molecular differences between primitive lung cancer and the metastatic site.

SUMMARY:
investigate the molecular differences between primitive lung cancer and the metastatic site.

ELIGIBILITY:
Inclusion Criteria:

* patients aged ≥18 years fit enough to tolerate the surgical operation;
* the operative risk is considered low based on respiratory reserve and cardiac assessment;
* the patient has clearly expressed willingness to adhere;
* availability of pathological material for tumor DNA extraction and NGS execution.

Exclusion Criteria:

* Women of childbearing age, pregnant or breastfeeding, or intending to become pregnant during the study.
* Any other illness, metabolic disorder, physical examination, or laboratory findings that constitute a contraindication to study participation.
* Recent or ongoing severe or clinically significant infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient diagnosed with NSCLC
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2025-12-18 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
To investigate the molecular differences between primitive lung cancer and the metastatic site. | From baseline to 18 months
  Tumoral DNA will be extracted from the formalin-fixed paraffin-embedded (FFPE) block containing the highest percentage of tumor cells, with macrodissection, if necessary, to obtain at least 30% of tumor cells. DNA was extracted from FFPE samples. Next-generation sequencing (NGS) analysis will be performed as previously described. Gene amplification is defined by a coverage mean superior to 3SD.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Spaggiari, Principal Investigator — European Institute of Oncology
Locations (1):
- Istituto Europeo di Oncologia, Milan, Italy